CLINICAL TRIAL: NCT04048720
Title: Norwalk Drop-In Family Nurture Intervention
Brief Title: Norwalk Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Norwalk Housing Authority (NHA) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAS0112
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Behavior Problem; Development Delay; Emotional Disturbances; Family Conflict; Relation, Mother-Child
Keywords: Family Nurture Intervention; Martha G. Welch MD; Feasibility Study; Preschool intervention; Co-regulation; Emotional Connection; Multiple Family Group Intervention
MeSH Terms: conditions — Mental Disorders; Learning Disabilities; Affective Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family Nurture Intervention (FNI) (Experimental): FNI sessions will be held once a week in the afternoon for eight weeks. Participants will take part in FNI group therapy with their child alongside other mother-child pairs. One to two staff members will lead FNI sessions.
  Interventions: Behavioral: Family Nurture Intervention

INTERVENTIONS:
Behavioral: Family Nurture Intervention — The mother-child pair will be asked to talk and play with each other as the pair customarily does. If the child becomes restless and dysregulated, the mother will be coached by the Nurture Specialist to bring the child back into a calm state through sustained physical contact, comforting touch, soothing words and eye contact. Each dyad will be offered eight group FNI sessions.
  Other Names: FNI

SUMMARY:
The purpose of this study is two-fold: 1) to examine the feasibility of the Drop-In model of Family Nurture Intervention (FNI); and 2) to collect pilot data concerning the mother's response to the Drop-In model of FNI and short term effects of participation. Feasibility of the Program will be measured through costs, staffing, space availability, and uptake. Participation in the Drop-In entails weekly visits for FNI. The investigators hypothesize that the Family Nurture Intervention will show feasibility through attendance and positive response to the Drop-In format. The investigators also expect the Family Nurture Intervention to improve mother's perceived well-being and mother-child emotional connection.

DETAILED DESCRIPTION:
Family Nurture Intervention (FNI) is a novel family-based program that facilitates mother-child emotional connection and co-regulation. Many current interventions aim at helping the child to self-regulate with or without the mother's help. However, the ability of the mother-child dyad to promote optimal development is dependent on their ability to co-regulate. The interactive co-regulation between the mother and the child shapes the behavior of both the mother and the child.

This study aims to investigate the feasibility and short term effects of participation in the Family Nurture Intervention for preschool aged children with developmental and behavior problems. Mothers and children will be engaged by Nurture Specialists in comforting and calming interactions to co-regulate with each other during weekly group sessions with the support of study staff. Intervention sessions will occur over the course of eight weeks, and each mother will decide how many sessions to attend.

ELIGIBILITY:
Inclusion Criteria:

* Mother is fluent in English or Spanish
* Mother is 18 years of age or older at the time of consent
* Mother-child pair does not demonstrate emotional connection as measured by the WECS
* Child is between the ages of 2 to 4½ years at date of enrollment (child must be younger than 4 years and 9 months at baseline assessment) or between 2 to 4½ at date of enrollment in study AAAQ9547
* Child resides with mother

Exclusion Criteria:

* The child has severe congenital anomalies or chromosomal anomalies including Downs syndrome and Cerebral Palsy
* The child has a diagnosis of Autism Spectrum Disorder
* The child has severe motor or physical disability
* Mother currently presents with psychosis or is currently taking antipsychotic medication
* Current maternal drug and/or alcohol abuse
* Mother is more than four months pregnant
* Mother and/or infant has a medical condition or contagion that precludes intervention components
* Mother is unable to commit to study schedule

Ages: 24 Months to 78 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Mother-child session interest | 8 weeks
  Study staff will track interest level and engagement with FNI through weekly forms and notes; mothers will be asked to give feedback on their experience of the study at the completion of eight weeks.
Change in videotaped Welch Lap Test | 8 weeks
  Mother-child 5-minute videotaped interactions, recorded weekly after each session, will be assessed for social engagement and emotional connection via the Welch Emotional Connection Screen (WECS).
  The Welch Emotional Connection Scale (WECS) construct is emotional connection between mother and child, which the investigators hypothesize predicts optimal development. There are four items on the WECS: Mutual Attraction, Mutual Vocal Exchange, Mutual Facial Engagement, and Mutual Sensitivity/Reciprocity. Each item is rated on a scale from 1 to 3 in 0.25 increments with a score of 3 considered optimal. There is also a binary question to the rater asking if the pair is emotionally connected - yes or no. The mother and child are scored as a pair, not individually.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Welch, MD, Principal Investigator — Columbia University
Locations (1):
- Norwalk Housing Authority, Norwalk, Connecticut, United States